CLINICAL TRIAL: NCT05246644
Title: Pilot Randomized Trial of Intravenous or Oral Acetaminophen After Cardiac Surgery
Brief Title: IV Acetaminophen After Cardiac Surgery - PILOT
Acronym: IVACS-Pilot
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Montreal Heart Institute (Other); University of Manitoba (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, magder sheldon, Senior Physician, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MUHC-ACETAMINOPHEN
Record Dates: First submitted 2021-12-15; First posted 2022-02-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: randomized double blind double dummy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: blinded medication with codes kept in the pharmacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Acetaminophen (Experimental): subjects will receive IV acetaminophen and a placebo oral acetaminophen starting immediately after surgery and for 8 doses
  Interventions: Drug: acetaminophen
- Oral acetaminophen (Active Comparator): subjects will receive a placebo for IV acetaminophen and active oral acetaminophen starting immediately after surgery and for 8 doses
  Interventions: Drug: acetaminophen

INTERVENTIONS:
Drug: acetaminophen — we will use IV acetaminophen and an oral placebo or IV placebo and active oral acetaminophen
  Other Names: placebo

SUMMARY:
Double blind double dummy of Intravenous Acetaminophen and oral acetaminophen placebo versus IV placebo versus oral acetaminophen in patients following cardiac surgery. The primary endpoint is development of Delirium during the post-operative stay.

DETAILED DESCRIPTION:
The study is randomized, double-blinded, and multicentre. Enrollment includes patients 18 years or older who are going for aortocoronary bypass surgery, single valve, or bypass and single valve. The intervention is blinded IV acetaminophen and blinded oral active or placebo acetaminophen . The study will start with a pilot trial of 120 patients at 4 centers- 30 at each site, 15 per group. The pilot is a vanguard. If the pilot shows appropriate compliance with the protocol, reliable blinding and appropriate enrolment, the results will not be unblinded but rolled into the full study. Stratification will be by site and age < 60 or >= 60.

ELIGIBILITY:
Inclusion Criteria:

* subjects > 18 years of age undergoing elective aortocoronary bypass, single valve replacement or single valve and aortocoronary bypass surgery

Exclusion Criteria:

* • Refusal by surgeon for inclusion of the patient

  * Requested late extubation by anesthesia or surgeon
  * Intra-aortic balloon pump
  * Sensitivity to acetaminophen
  * Pre-operative cognitive dysfunction
  * Psychiatric history with active treatment
  * Parkinson's disease
  * Alzheimer's disease
  * Medication for cognitive decline
  * History of recent seizures
  * Recent history of alcohol misuse
  * Creatinine clearance less than 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Development of delirium post operatively | up to 7 days post operatively
  Incidence of delirium will be analyzed between patients treated with IV or oral acetaminophen, measured from 24 hours post-operation and daily until discharge. Delirium will be defined as an acute change in pre-operative baseline condition with additional features of inattention and either disorganized thinking and altered loss of consciousness, as defined by the Confusion Assessment Method (CAM) or CAMICU when in the intensive care unit

SECONDARY OUTCOMES:
total opioid usage | up to 7 days post-operatively
  tabulation of all opioids normalized to morphine
Numeric pain rating scale | up to 48 hours
  visual pain score from 1 to 10
cognitive function | 7 days post-operative, 6 months and 1 year
  change in cognitive function score by 2 based on the Montreal cognitive assessment
hospital length of stay | length of stay is measured from the day of surgery until the day of discharge from hospital in days
  Days until discharge
Intensive care length of stay | ICU stay is measured from the hour of arrival in the ICU and until the patient leaves the ICU in hours
  hours in ICU

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec